CLINICAL TRIAL: NCT06216509
Title: Endoscopic Ultrasound-Guided Portosystemic Pressure Gradient Measurements in Patients with Cirrhosis and Non Cirrhotic Portal Hypertension
Brief Title: Endoscopic Ultrasound-Guided Portosystemic Pressure Gradient Measurements
Acronym: EUSPREM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Collaborators: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Andrada Seicean, Clinical Professor, Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 187214022023
Record Dates: First submitted 2023-02-16; First posted 2024-01-22 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis; Vascular Diseases
Keywords: portal pressure gradient; endoscopic ultrasound; HVPG; portal hypertension
MeSH Terms: conditions — Fibrosis; Vascular Diseases; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cirrhosis (Other): patients with cirrhosis undergoing TIPS placement
  Interventions: Device: Endoscopic ultrasound pressure measurement
- porto sinusoidal vascular disorder and portal vein thrombosis (Other): patients with porto sinusoidal vascular disorder and portal vein thrombosis either in the context of cirrhosis or non cirrhotic portal vein thrombosis
  Interventions: Device: Endoscopic ultrasound pressure measurement

INTERVENTIONS:
Device: Endoscopic ultrasound pressure measurement — all eligible patients from both groups will undergo Endoscopic ultrasound pressure measurement under sedation.

SUMMARY:
Portal hypertension (PHT) is the main consequence of advanced chronic liver diseases (ACLD) and is often associated with severe complications leading to increased morbidity and mortality. Currently, the gold standard for the evaluation of the severity of PHT is the hepatic venous-pressure gradient (HVPG). The disadvantage of using the HVPG, besides the availability of the technique only in referral centres, is in the case of patients with vascular liver disorders because the HVPG underestimates the severity of PHT. Recent studies have evaluated the feasibility of the pressure gradient measurement through endoscopic transgastric and transhepatic access using special kit with a 25-gauge FNA needle (Cook Medical, Winston-Salem, NC, USA) and a compact manometer (Cook Medical, Bloomington, Ind, USA) that has the disadvantage of high purchase cost, no tracing of pressure possible and has not yet been properly correlated with the gold standard HVPG measurement or PPG measurement thus limiting its use in current practice. The aim of the study is 1. to assess and compare the correlations in the porto-systemic gradient measurement between a) direct portal vein puncture during TIPS insertion, b) direct portal and hepatic pressure measurements using a 22 Gauge FNA needle during endoscopic ultrasound procedure and c) indirect portal vein pressure measurements using the interventional radiology based hepatic HVPG procedure in patients with cirrhosis submitted to TIPS procedure for complications of portal hypertension and 2. To evaluate and compare the porto-systemic gradient obtained by direct portal and hepatic pressure measurements using a 22 Gauge FNA needle during endoscopic ultrasound and indirect measurement through HVPG measuring in patients with presinusoidal hypertension and those with portal vein thrombosis.

DETAILED DESCRIPTION:
Number of patients needed to be included:

To achieve the first primary objective, the investigators will include 20 patients. To achieve the second primary objective, 30 patients will be included, with presinusoidal portal hypertension and patients with non-cirrhotic portal vein thrombosis or portal vein thrombosis in the context of cirrhosis. As non-cirrhotic portal hypertension is a lesser frequent type of portal hypertension, the number needed to be included will be sufficient.

Duration of the Study and Patient Participation:

Patient enrolment is expected to be completed within 24 months of study initiation. Total study duration is expected to be 26 months. Patients are expected to participate in this study for 7 days after the study procedure. Patients who meet one or more exclusion criteria during evaluation with EUS will be followed through procedural timepoint.

Patient Consent Patients who meet the inclusion criterion and none of the exclusion criteria will be invited to participate in this study. Patients eligible for enrolment will have the clinical study explained to them and each patient who agrees to participate will sign and date an informed consent document prior to the procedure or any study-specific testing or assessments.

Methods:

1. Patient Screening- Review inclusion criteria and exclusion criteria;Review study with the patient and obtain written informed consent; Record medication and laboratory tests
2. Day of the study 2.1. Patients with cirrhosis undergoing TIPS placement and indication for varices assessment: In this study the investigators will correlate the PPG obtained by direct portal and hepatic pressure measurements using a 22 Gauge FNA needle during endoscopic ultrasound procedure for varices assessment and indirect portal vein pressure measurements using the interventional radiology based hepatic HVPG procedure in patients with cirrhosis under general anaesthesia.

A. General anesthesia B. HVPG measurements will begin prior to TIPS procedure. Before the TIPS placement, standard HVPG measurement will be performed according to the practice standard of care after administration of broad-spectrum prophylactic antibiotics 1 hour prior to procedure. Briefly, the patients will be placed in the angiography room in supine position and the '0' from the arterial pressure measurement kit will be placed at the mid axillary line and pressures will be zeroed. Then, under ultrasound guidance, the right internal jugular vein will be catheterized with a 10 Fr introducer. Thereafter, with a 7Fr balloon-occluded catheter, the right atrium and the inferior retrohepatic vena cava pressures will be recorded. Using the same catheter, the right or the middle suprahepatic vein will be catheterised and 2 ml of iodine contrast will be injected to ensure adequate occlusion after inflation of the balloon. If collaterals are present, they will be recorded. The wedge pressure (WHVP) will be measured in triplicate and, after 1min and 30 seconds and until stabilization, the pressures will be recorded. The free hepatic venous pressure (FHVP) will be measured at the level of the IVC ostium.

C. Direct FHVP and Portal pressure measurement during EUS procedure. Using EUS guidance, assessment of esophageal and/or gastric varices will be performed, as indicated for each case. The patients will be evaluated for possible local direct puncture contraindications. If no contraindications will be found, the free hepatic vein pressure and portal pressure will be measured through direct puncture of the vessels, left or medial hepatic vein and portal vein, respectively. The puncture will use a 22 G FNA Needle and 1 ml of heparinized saline will be flushed to confirm the good puncture location. Thereafter, the needle will be connected to the hemodynamic pressure measurement kit and the pressures will be recorded D. Direct portal pressure measurement during TIPS procedure. The portal pressure will be measured after the direct puncture of the portal vein during TIPS procedure before angioplasty and stent placement. Thereafter, the TIPS procedure will proceed as standard of care.

2.2.Study 2. Patients with presinusoidal portal hypertension or portal vein thrombosis: In this study the investigators will assess the correlation of the PPG obtained by direct portal and hepatic pressure measurements using a 22 Gauge FNA needle during endoscopic ultrasound under mild sedation procedure and portal hypertension signs in patients with presinusoidal portal hypertension and those with cirrhotic or non-cirrhotic portal vein thrombosis.

A. Patients will undergo HVPG measurement under no sedation B. Direct FHVP and Portal pressure measurement during EUS procedure as outlined above will be performed under mild sedation

All measured pressures will be recorded as source documentation and will be reviewed by an independent physician for quality with vast experience in HVPG pressure tracings

Follow-up: same day of the procedure; at 24-48 hours; at 1 week- assessment of complications

Safety Reporting:

All adverse events and device deficiencies identified by the investigator as being relevant to any of the procedures (e.g. HVPG, TIPS, EUS procedure) that occur after the point of enrolment until the last day of patient participation up to 7 days after the study procedure, will be reported by the investigators in special CRFs.

ELIGIBILITY:
Inclusion Criteria:

patients with cirrhosis undergoing TIPS placement and patients with presinusoidal portal hypertension and patients with portal vein thrombosis

Exclusion Criteria:

1. Patient is < 18 or > 85 years of age
2. Patient is pregnant, breast-feeding, or planning to become pregnant during the course of the study
3. Patient is unwilling or unable to sign and date the informed consent
4. Patient for whom endoscopic procedures are contraindicated
5. Patients for whom propofol general anesthesia is contraindicated
6. Previous transjugular intrahepatic or surgical portosystemic shunt
7. Previous total or partial splenectomy
8. Known history of spontaneous bacterial peritonitis (SBP) within the last three months irrespective of treatment for SBP
9. Patients with known infection which is not controlled by medical intervention
10. Severe Portopulmonary hypertension contraindicating TIPS placement
11. Cardiac decompensation
12. Cholestatic liver disease
13. Patients with current advanced hepatocellular carcinoma (HCC)
14. Emergent salvage TIPS placement in patients with failure to control bleeding
15. Severe coagulopathy
16. Anatomic abnormalities of the hepatic vasculature that prevent access to the intrahepatic portion of the portal vein or hepatic veins
17. Evidence of active gastrointestinal bleeding
18. If the volume of ascites in the path of the needle prevents apposition of the gastrointestinal tract and liver
19. Allergies to iodine contrast

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Correlation of the porto systemic pressure gradient measured by EUS and TIPS | 1 year
  in the first 12 months, patients enrolled will perform EUS and TIPS placement; measurement will be done according to protocol
Correlation of the hepatic venous pressure gradient and portosystemic pressure gradient | 1 year
  in the first 12 month, patients enrolled will perform EUS and TIPS placement; measurement will be done according to protocol
Correlation of the porto systemic pressure gradient and portal hypertension signs | 1 year
  in the next 12 months, patients meeting criteria will perform EUS pressure assessment and detection of varices

CONTACTS AND LOCATIONS:
Overall Officials: Andrada Seicean, Prof MD PhD, Principal Investigator — Institutul Regional de Gastroenterologie si Hepatologie Prof Dr Octavian Fodor
Locations (1):
- Regional Institute of Gastroenterology and Hepatology Prof. Dr. O. Fodor, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Samarasena JB, Huang JY, Tsujino T, Thieu D, Yu A, Hu KQ, Lee J, Chang KJ. EUS-guided portal pressure gradient measurement with a simple novel device: a human pilot study. VideoGIE. 2018 Oct 25;3(11):361-363. doi: 10.1016/j.vgie.2018.07.013. eCollection 2018 Nov. PMID 30402586
- [Background] Huang JY, Samarasena JB, Tsujino T, Chang KJ. EUS-guided portal pressure gradient measurement with a novel 25-gauge needle device versus standard transjugular approach: a comparison animal study. Gastrointest Endosc. 2016 Aug;84(2):358-62. doi: 10.1016/j.gie.2016.02.032. Epub 2016 Mar 3. PMID 26945557